CLINICAL TRIAL: NCT05115318
Title: The Effect of Medical Cannabis on Tics, Premonitory Urge and Psychiatric Comorbidity in Adults With Tourette Syndrome
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0491-10-TLV
Record Dates: First submitted 2021-10-16; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Tourette Syndrome; Cannabis
Keywords: Cannabidiol; Cannabis; Medical Cannabis; delta(9)-Tetrahydrocannabinol; Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome; Marijuana Abuse | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Tourette syndrome patients: Patients will be assessed before (baseline), 4 (visit 2) and 12 weeks (visit 3) after use of Medical cannabis via inhaled dried buds or sublingual oil extract. The percentage of THC and CBD were pre-set to 10% and 2%, respectively. All patients received the same general instructions for treatment titration, which was to start with 1 drop or puff a day and increase by 1 drop or puff as needed. There was no fixed schedule for the incremental increases, thus each patient freely raised the dose as well as number of daily consumptions until clinical benefit was achieved or SE emerged over a follow-up period of 12 weeks.
  Interventions: Drug: Medical Cannabis

INTERVENTIONS:
Drug: Medical Cannabis — Patients with GTS were assessed before, 4 and 12 weeks after Medical cannabis initiation for consumption habits, efficacy and side effect profile

SUMMARY:
Medical cannabis (MC) is a standard treatment in Israel to adults with resistant Gilles de la Tourette syndrome (GTS). While small randomized control trials assessed THC efficacy on tics and premonitory urge, only small retrospective studies assessed MC efficacy and tolerability in GTS. Herein, By using an open-label, prospective design, our aim is to determine the preferred method of use, efficacy and tolerability of 12 weeks of treatment with MC in adult patients with GTS.

DETAILED DESCRIPTION:
Gilles de la Tourette syndrome (GTS) is a childhood onset neuropsychiatric disorder characterized by the presence of multiple motor and one or more phonic tics continuing for at least one year. In Israel, although consumption of cannabis is outlawed, there is an option to allow patients to consume the drug under supervision. Medical Cannabis (MC) consumed by inhalation of smoked or vaporized dried female buds, or subligual oil extract of whole plant, has been an approved treatment by the Ministry of Health (MOH) for resistant GTS since 2013. Previous studies suggested that MC has a good effect on tics, quality of like and with good tolerability among patients with resistant GTS.

In the current study, we prospectively followed-up patients eligible for MC according to MOH restrictions, at our GTS clinic at the Tel-Aviv Sourasky Movement Disorders Unit (MDU). Each subject signed a written informed consent before inclusion in the trial. Also, since driving under the influence of cannabis is forbidden by the Israeli law, patients were instructed and gave their oral commitment to avoid driving. The study was approved by the research ethics (Helsinki) committee at our center. MC was consumed as oil extract, vaporized, or smoked dried buds. The treating neurologist (S.A.) and patient together decided on the method of consumption during the visit before initiating treatment. Patients were assessed 4 and 12-weeks following treatment initiation to gather data regarding treatment efficacy, tolerability and SEs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Diagnosis of GTS confirmed by the treating neurologist based on the DSM-V criteria
* Eligibility to receive MOH MC license for GTS
* Provided written informed consent

Exclusion Criteria:

* Regularly use cannabis in any form for self-medication prior to entering the study
* Pregnant or lactating women
* Have a tic disorder other than GTS
* Have concurrent physical or mental disease that could interfere with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with resistant Tourette syndrome
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in vocal and motor tics and disease burden | Baseline, after 4 and 12 weeks since treatment initiation
  Using Yale Global Tic Severity Scale (YGTSS), range 0-100, higher scores mean a worse outcome
Change in premonitory urge | Baseline, after 4 and 12 weeks since treatment initiation
  using Premonitory Urge for Tic Scale (PUTS), range 0-36, higher scores mean a worse outcome
Subjective improvement of tics and Quality of life | Baseline, after 4 and 12 weeks since treatment initiation
  Using a 7-point Likert-type scale, range 1-7, higher scores mean a better outcome

SECONDARY OUTCOMES:
Examine patient's tetrahydrocannabinol-9-delta (THC) and Cannabidiol (CBD) consumption per month | After 12 weeks since treatment initiation
  Measuring total THC and CBD consumption per month in grams
Assessment of major side effects of treatment | After 4 and 12 weeks since treatment initiation
  report (yes/no) on side effects from list and (free text) to add notes on side effect. List: Anxiety, Cognitive, Dizziness, Sedation, Fatigue, Red eyes
  , Dry mouth, Gastrointestinal

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No